CLINICAL TRIAL: NCT03152149
Title: INvestigating COPD Outcomes, Genomics and Neutrophilic Inflammation With Tiotropium and Olodaterol
Acronym: INCOGNITO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Boehringer Ingelheim (Industry); NHS Tayside (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2016RC22; 2016-004473-41 (EudraCT Number)
Record Dates: First submitted 2017-05-01; First posted 2017-05-12 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tiotropium-olodaterol; fluticasone furoate; vilanterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. Spiolto Respimat (Active Comparator): Spiolto Respimat (Tiotropium 2.5 micrograms,olodaterol 2.5 micrograms) 2 puffs once daily for 6 months
  Interventions: Drug: Tiotropium & olodaterol
- 2. Relvar Ellipta (Active Comparator): Relvar Ellipta (fluticasone furoate 92 micrograms, vilanterol 22 micrograms) 1 puff once per day for 6 months
  Interventions: Drug: fluticasone furoate & vilanterol

INTERVENTIONS:
Drug: Tiotropium & olodaterol — Spiolto Respimat (Tiotropium 2.5 micrograms,olodaterol 2.5 micrograms) 2 puffs once daily for 6 months
  Other Names: Spiolto Respimat
  Arms: 1. Spiolto Respimat
Drug: fluticasone furoate & vilanterol — Relvar Ellipta (fluticasone furoate 92 micrograms, vilanterol 22 micrograms) 1 puff once per day for 6 months
  Other Names: Relvar Ellipta
  Arms: 2. Relvar Ellipta

SUMMARY:
This protocol describes a randomised controlled trial to test the hypothesis that 6 months of treatment with tiotropium and olodaterol will result in a reduction in bacterial load, an improvement in neutrophilic inflammation and clinical benefits compared with treatment with inhaled fluticasone furoate and vilanterol in patients with neutrophilic Chronic obstructive pulmonary disease (COPD).

COPD is the third leading cause of death worldwide and a major cause of morbidity in the UK. Exacerbations drive disease progression and worsening quality of life and therefore prevention of exacerbations has been a major goal of treatment.

In recent years, attempts have been made to phenotype COPD patients in order to target therapies to the correct groups of patients that will benefit. Inhaled corticosteroids (ICS) are primarily effective for patients with eosinophilic inflammation, while there are few established therapies for patients with neutrophilic disease. In recent years, all ICS preparations have been associated with a significant increased risk of pneumonia and this risk appears to be greatest in patients with non-eosinophilic inflammation. Combined treatment with long acting beta-agonists (LABA) and long acting muscarinic antagonists (LAMA) combinations appears to be a safer and more effective alternative for patients with non-eosinophilic disease. The combination of tiotropium and olodaterol in particular, has strong preclinical data supporting beneficial effects on neutrophilic inflammation.

The trial is a multi-centre randomised open label controlled parallel group study with two treatment arms in 80 participants. Moderate to very severe COPD patients and currently treated with inhaled corticosteroid therapy will be randomised to treatment with either the combination of tiotropium and olodaterol (LABA/LAMA) or fluticasone furoate and vilanterol (ICS/LABA). Participants will return at 1 month, 2 months, 3 months and 6 months for sampling of the lower airway by sputum samples and the upper airway using oropharyngeal and nasopharyngeal swabs. Sputum will be used to test for airway neutrophilic inflammation.

This study will make an important contribution to understanding "phenotyping" in COPD by identifying whether the combination of tiotropium and olodaterol improves airway bacterial load and restores neutrophil function in patients with neutrophilic COPD.

DETAILED DESCRIPTION:
BACKGROUND Inhaled corticosteroids (ICS) are commonly prescribed for patients with chronic obstructive pulmonary disease (COPD), but their role in the management of COPD is currently being re-evaluated in light of new evidence and the emergence of alternative treatments. Recent concerns have been expressed about the safety of ICS in COPD following several randomized controlled trials of fluticasone propionate and fluticasone furoate demonstrating an increase in rates of pneumonia as an adverse event. Several systematic reviews and observational studies confirm an association between ICS use and risk of pneumonia.

A series of post-hoc analyses of large randomized controlled trials of ICS/ long acting beta-agonists (LABA) or ICS alone have suggested that benefits of ICS in terms of exacerbation reduction and preventing lung function decline are limited to a subgroup of patients with eosinophilic airway inflammation. Eosinophils are highly sensitive to ICS, and so there is a compelling rationale for this association, and therefore an emerging consensus that ICS should be reserved for those patients with eosinophilic disease. This can be identified on the basis of blood eosinophil count although the precise cut-off is yet to be determined. This is strongly supported by a post-hoc analysis of the WISDOM randomized controlled trial of ICS withdrawal in which ICS withdrawal was only associated with an increase in exacerbations above blood eosinophil counts of 300 cells per ul. Furthermore in the FLAME study which excluded patients with very high eosinophils counts, LABA/long acting muscarinic antagonists (LAMA) was superior to ICS/LABA in terms of reducing exacerbations.

If there is an emerging consensus regarding the treatment of "eosinophilic COPD", then the unmet need in the management of COPD is for the majority of patients that have neutrophilic airway inflammation. Neutrophilic inflammation does not respond to inhaled corticosteroids and indeed there is in-vitro evidence that inhaled corticosteroids may exacerbate neutrophilic inflammation by delaying neutrophil apoptosis. Neutrophilic inflammation is associated with disordering of the lung microbiome with overgrowth of Proteobacteria, a process that may be exacerbated by ICS. Release of proteolytic enzymes such as elastase and matrix metalloproteinase from neutrophils are associated with disease progression and lung function decline in COPD.

RATIONALE FOR STUDY It is hypothesised that the combination of tiotropium and olodaterol may be an ideal treatment option for patients with neutrophilic COPD because

* Tiotropium and olodaterol have both been shown to have potentially beneficial effects in suppressing neutrophilic inflammation without impairing bacterial killing
* These effects may reverse the detrimental impact of inhaled corticosteroids on airway neutrophil function and the microbiome.

In particular olodaterol was evaluated in cigarette smoke- and Lipolpolysaccharide - induced- models of neutrophil lung inflammation in mice and guinea pigs. The results showed Olodaterol to suppress neutrophil recruitment to the lung (by up to 90%) while preserving chemotactic function (which is required for effective phagocytosis of pathogens). Tiotropium has also been extensively investigated and is known to suppress neutrophil recruitment and neutrophil dependent remodelling in a number of in-vivo models and may work synergistically with olodaterol in reducing neutrophil retention in the lung.

This extensive preclinical work justifies a study of olodaterol/tiotropium in human subjects evaluating its impact on neutrophilic inflammation. This could establish the combination of olodaterol/tiotropium as the first line therapy for patients with neutrophilic COPD.

This trial will compare treatment of patients with COPD previously treated with ICS randomized to either tiotropium/olodaterol combination or fluticasone furoate/vilanterol combination. The objective of the trial is to evaluate in-vivo effects of these drugs on the lung microbiota and airway neutrophil function. In particular, we expect that 6 months treatment with olodaterol/tiotropium will result in a reduced airway bacterial load (through restored neutrophil function allowing neutrophils to kill airway bacteria), an increase in microbiota diversity, an enhanced ex-vivo killing of Haemophilus influenzae and reduced markers of neutrophilic airway inflammation.

HYPOTHESIS Tiotropium and olodaterol combination treatment will result in a reduced airway bacterial load at 6 months compared to fluticasone furoate and vilanterol. The reduced bacterial load will be associated with improvements in the airway microbiota and reduced markers of neutrophilic inflammation and restored neutrophil function.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged > 40 years
* Current or ex-smokers having at least a 10 pack year smoking history
* A clinical diagnosis of Chronic Obstructive Pulmonary Disease (COPD) made by a physician
* Post-bronchodilator Forced Expiratory Volume 1 (FEV1)/Forced Vital Capacity ratio at screening of <70%
* Moderate to Very Severe COPD (GOLD II-IV) according to consensus guidelines consisting of a post-bronchodilator FEV1 <80% predicted at screening.
* Currently treated with inhaled corticosteroids (with or without long acting bronchodilators) for at least 12 months prior to screening.
* Able to perform all study procedures including spirometry and questionnaires with minimal assistance
* Blood eosinophil count less than 300 eosinophil cells per microlitre on bloods taken at screening.
* Able to produce a sputum sample at the baseline visit (either spontaneously or with nebulised saline induction)

Exclusion Criteria:

* Inability to give informed consent
* Asthma
* Acute Antibiotics within 28 days prior to screening
* Long term macrolide therapy if newly commenced in the past 3 months
* Current use of the following: roflumilast, ritonavir, itraconazole, telithromycin, or ketoconazole (or other strong CYP3A4 inhibitors).
* Systemic Immunosuppressive medication including current oral corticosteroids at a dose >5mg for >28 days.
* Glomerular filtration rate (eGFR) below 30ml/min/1.73m2 or requiring dialysis. This will be determined at screening.
* Use of any investigational drugs within five times of the elimination half-life after the last study dose or within 30 days, whichever is longer.
* Known allergy, intolerance or contraindication to any of the study drugs
* Unstable co-morbidities (cardiovascular disease, active malignancy) which in the opinion of the investigator would make the patient unsuitable to be enrolled in the study
* An exacerbation of COPD occurring during the 28 days prior to screening requiring treatment with either oral corticosteroids or antibiotics.
* An exacerbation requiring treatment with antibiotics or corticosteroids between the screening and randomization visit
* Pregnancy or breast feeding
* Women of child bearing potential who are not practicing an acceptable method of contraception
* Long term oxygen therapy
* Lapp lactase deficiency, glucose-galactose malabsorption or another inherited disorder of galactose metabolism.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Change in bacterial load of total bacteria determined by quantitative polymerase chain reaction | From baseline to 1, 2, 3 and 6 months
  To determine the effects of the Tiotropium and olodaterol combination vs fluticasone furoate and vilanterol on airway bacterial load from sputum

SECONDARY OUTCOMES:
Change in bacterial community composition determined by 16S microbiome sequencing as measured by the Shannon Diversity index. | From baseline to 1, 2, 3 and 6 months
  To determine the effects of the Tiotropium and olodaterol combination vs fluticasone furoate and vilanterol on the airway microbiota. Microbiota will be characterised in sputum, oropharyngeal swabs and nasopharyngeal swabs
Sputum neutrophil elastase activity determined using an activity based immunoassay | From baseline to 1, 2, 3 and 6 months
  To determine the effects of the Tiotropium and olodaterol combination vs fluticasone furoate and vilanterol on sputum neutrophil elastase activity
Change in sputum neutrophil extracellular traps determined using a validated ELISA | From baseline to 1, 2, 3 and 6 months
  To determine the effects of the Tiotropium and olodaterol combination vs fluticasone furoate and vilanterol on concentration sputum neutrophil extracellular traps
Change in sputum cytokines and inflammatory markers including but not limited to CXCL-8, IL17, IL-1beta, resistin, IL13 | From baseline to 1, 2, 3 and 6 months
  To determine the effects of the Tiotropium and olodaterol combination vs fluticasone furoate and vilanterol on sputum cytokines and inflammatory markers

OTHER OUTCOMES:
Relative abundance of Haemophilus Operational Taxonomic Units at genus level or relative abundance of proteobacteria at phylum level. | Baseline, 1, 2, 3 and 6 months
  To determine the effects of the Tiotropium and olodaterol combination vs fluticasone furoate and vilanterol on the airway microbiota. Microbiota will be characterised in sputum, oropharyngeal swabs and nasopharyngeal swabs
Proportion of patients with dysbiosis as defined by >40% relative Operational Taxonomic Units of a single organism. | Baseline, 1, 2, 3 and 6 months
  To determine the effects of the Tiotropium and olodaterol combination vs fluticasone furoate and vilanterol on the airway microbiota. Microbiota will be characterised in sputum, oropharyngeal swabs and nasopharyngeal swabs
Comparison of adverse events/serious adverse events between groups on dual bronchodilators and inhaled corticosteroids | Baseline, 1, 2, 3 and 6 months
  To evaluate the safety and tolerability of Tiotropium and olodaterol combination vs fluticasone furoate and vilanterol in patients previously treated with inhaled corticosteroids
Bacterial community composition determined by 16s microbiome sequencing. | From baseline to 1, 2, 3 and 6 months
  To provide a longitudinal characterisation of the upper and lower airway microbiota in oropharyngeal/nasopharyngeal swabs and sputum in COPD
Mean fluorescence intensity by flow cytometry | From baseline to 1, 2, 3 and 6 months
  To determine the effects of the Tiotropium and olodaterol combination vs fluticasone furoate and vilanterol on neutrophil receptor expression - specifically expression of CD88, CD35, CD11b and CD41a in COPD patients
Change in ex-vivo phagocytosis of Haemophilus tested by incubating sputum cells with FITC-labelled H. influenzae | From baseline to 1, 2, 3 and 6 months
  To determine the effects of the Tiotropium and olodaterol combination vs fluticasone furoate and vilanterol on sputum neutrophil phagocytosis of Haemophilus influenzae
Quality of life St. George's Respiratory Questionnaire(SGRQ) | From baseline to 1, 2, 3 and 6 months
  To evaluate patient reported outcome measures between the groups treated with Tiotropium and olodaterol combination vs fluticasone furoate and vilantero using COPD assessment test (CAT)
Quality of life COPD assessment test (CAT) | From baseline to 1, 2, 3 and 6 months
  To evaluate patient reported outcome measures between the groups treated with Tiotropium and olodaterol combination vs fluticasone furoate and vilantero using MRC dyspnoea score
Quality of life MRC dyspnoea score | From baseline to 1, 2, 3 and 6 months
  To evaluate patient reported outcome measures between the groups treated with Tiotropium and olodaterol combination vs fluticasone furoate and vilantero using St. George's Respiratory Questionnaire(SGRQ)
Quality of life transitional dyspnoea index | From baseline to 1, 2, 3 and 6 months
  To evaluate patient reported outcome measures between the groups treated with Tiotropium and olodaterol combination vs fluticasone furoate and vilantero using the transitional dyspnoea index
Comparison of time to first exacerbation of Chronic Obstructive Pulmonary Disease | From baseline to 1, 2, 3 and 6 months
  To evaluate if changes in the airway microbiota or airway inflammatory profiles are associated with time to first exacerbation of Chronic Obstructive Pulmonary Disease
Number of exacerbations of Chronic Obstructive Pulmonary Disease | From baseline to 1, 2, 3 and 6 months
  To evaluate if changes in the airway microbiota or airway inflammatory profiles are associated with number of exacerbations of Chronic Obstructive Pulmonary Disease
Change in FEV1 | From baseline to 1, 2, 3 and 6 months
  To evaluate if changes in the airway microbiota or airway inflammatory profiles are associated with change in FEV1

CONTACTS AND LOCATIONS:
Overall Officials: James Chalmers, MBChB, MRCP, Principal Investigator — University of Dundee
Locations (4):
- United Kingdom (4):
  - NHS Tayside, Dundee
  - NHS Greater Glasgow and Clyde, Glasgow
  - Northumbria Healthcare NHS Foundation Trust, North Shields
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: Undecided